CLINICAL TRIAL: NCT00006066
Title: Phase I/II Trial of Subcutaneous IL-2 With Highly Active Antiretroviral Therapy in HIV-Infected Children With Immunosuppression
Brief Title: Interleukin-2 Plus Anti-HIV Therapy in HIV-Infected Children With Weakened Immune Systems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 402; 10607 (Registry Identifier: DAIDS ES Registry Number); PACTG 402
Record Dates: First submitted 2000-07-14; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Injections, Subcutaneous; Interleukin-2; Dose-Response Relationship, Drug; Drug Therapy, Combination; Immunocompromised Host; CD4 Lymphocyte Count; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Tetanus Toxoid; J protein, Bacteriophage phi X 174; aldesleukin

INTERVENTIONS:
Biological: Diphtheria & Tetanus Toxoids & Acellular Pertussis Vaccine Adsorbed
Biological: Diphtheria and Tetanus Toxoids Adsorbed
Biological: Tetanus and Diphtheria Toxoids Adsorbed
Drug: Bacteriophage phi X 174
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to determine the safety of a drug called interleukin-2 (IL-2) given with anti-HIV therapy in children with HIV infection. This study will also determine the best dose of IL-2 to give children.

IL-2 is an important substance produced by the body's white blood cells that helps the body fight infection. People with HIV infection do not produce enough IL-2. It is hoped that IL-2 treatment will help boost the immune system in people with HIV infection. It has not been studied very much in children and doctors need to know what doses are safe to give.

DETAILED DESCRIPTION:
One of the challenges in effective combination therapy in HIV-infected patients is the ability to achieve immune reconstitution. IL-2 is hypothesized to restore and/or preserve the immune system when added to potent antiretroviral regimens. This study will evaluate restoration of immune functions of CD4 cells and will also determine the best way to deliver IL-2 in a safe and effective way.

Part I: Patients add a 5-day course of subcutaneous IL-2 every 8 weeks for up to 48 weeks (6 cycles) to their HAART therapy. Three dose levels of IL-2 are administered. [AS PER AMENDMENT 5/3/01: It is strongly recommended, but not required, that] the first and second cycles of IL-2 are given in the hospital on an inpatient basis. The parent or patient is trained to give the injections and has the option of administering subsequent injections at home. Patients are monitored for CD4 and CD8 cell count and viral load. Enrollment into Part 1 begins at the lowest dose level; assuming no serious toxicities (Grade 3 or higher) occur, patients are enrolled into higher dose levels. The highest tolerated dose is established.

Part 2: After the highest tolerated dose is established in Part 1, additional patients are randomized to receive HAART alone (Arm 1), HAART with high-dose IL-2 (Arm 2), or HAART with low-dose IL-2 (Arm 3). High-dose IL-2 is given twice daily at the highest dose tolerated in Part 1 for 5 days every 8 weeks for 6 cycles. Low-dose IL-2 is given once a day every day for 48 weeks. For Arms 2 and 3 [AS PER AMENDMENT 5/3/01: (except patients in the pharmacokinetic substudy), it is strongly recommended, but not required, that] IL-2 is given the first week on an inpatient basis by hospital personnel. As in Part 1, there is the option of administering the remaining injections at home. Intensive toxicity monitoring, routine lymphocyte subsets, and quantitative HIV RNA are performed on all patients at specified time points during the study. The first 12 patients in Arms 2 and 3 have pharmacokinetic testing with frequent blood samples drawn at intervals, some of which require staying up to 12 hours at the clinic. Diphtheria/tetanus immunizations and bacteriophage phi X174 immunizations are administered to all patients to determine antibody responses.

ELIGIBILITY:
Inclusion Criteria

A child may be eligible for this trial if he/she:

* Is HIV-positive.
* Is 2 to 18 years old (consent of parent or guardian required if under 18).
* Has received 12 or more weeks of anti-HIV drug therapy, consisting of at least 3 drugs. This combination may include a nucleoside reverse transcriptase inhibitor (NRTI), a nonnucleoside reverse transcriptase inhibitor, or a protease inhibitor, or 3 NRTIs. Combinations of NRTIs may not include abacavir (ABC). Patients may have taken ABC if it was not in combination with 2 other NRTIs. (This reflects a change in the requirement for anti-HIV therapy.)
* Has a plasma HIV RNA level of less than 10,000 copies/ml.
* Has evidence of a weakened immune system (based on CD4 cell counts and absolute CD4 percentage less than 25 percent). (This reflects a change in how a weakened immune system is defined.)
* Has a parent or guardian who is willing to comply with study requirements.
* Has symptoms of HIV infection.

Exclusion Criteria

A child will not be eligible for this study if he/she:

* Has an active opportunistic (AIDS-related) infection.
* Is pregnant.
* Is taking certain medications, such as steroids or other drugs that affect the immune system, within 6 weeks prior to study entry.
* Is taking ABC.
* Is taking certain antibodies.
* (Exclusion criteria reflect changes.)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92
Dates: Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Savita Pahwa, Study Chair
Locations (14):
- United States (13):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
- Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan, Puerto Rico